CLINICAL TRIAL: NCT01782950
Title: Evaluation of the Pharmacokinetics of Antituberculosis Drugs and Tuberculosis Treatment Outcomes in HIV-tuberculosis Co-infected Ugandan Adults
Brief Title: Evaluation of the Pharmacokinetics of Antituberculosis Drugs and Tuberculosis Treatment Outcomes
Acronym: SOUTH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Responsible Party: Principal Investigator, Infectious Diseases Institute, Principal Investigator, Makerere University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDI
Record Dates: First submitted 2013-01-09; First posted 2013-02-04 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: AIDS With Tuberculosis
Keywords: HIV; Tuberculosis; Antituberculosis drugs
MeSH Terms: conditions — Tuberculosis | interventions — Rifampin; Isoniazid; Ethambutol; Pyrazinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anti-tuberculosis drugs (Other): Rifampicin, Isoniazid, Ethambutol, Pyrazinamide tablets 3 to 5 tablets once daily for 2 months followed by Rifampicin, Isoniazid 3 to 5 tablets once daily for 4 months
  Interventions: Drug: Rifampicin, Isoniazid, Ethambutol, Pyrazinamide

INTERVENTIONS:
Drug: Rifampicin, Isoniazid, Ethambutol, Pyrazinamide — Rifampicin, Isoniazid, Ethambutol, Pyrazinamide: 3, 4 or 5 tablets daily for weight below 55kg, above 55kg or above 70kg respectively for first 2 months followed by Rifampicin, Isoniazid: 3, 4 or 5 tablets daily for patients' weight below 55kg, above 55kg or above 70kg respectively for 4 months
  Other Names: Forecox Trac; and Montozid

SUMMARY:
Tuberculosis (TB) is a leading cause of death in HIV-infected individuals. There are insufficient data correlating concentrations of anti-TB drugs with treatment response. We hypothesize that sub-therapeutic concentrations of anti-TB drugs are associated with inadequate TB treatment response to Mycobacterium tuberculosis.

DETAILED DESCRIPTION:
During the study periodic monitoring will be conducted to ensure that the protocol and Good Clinical Practices (GCPs) are being followed.The monitors may review source documents to confirm that the data recorded on CRFs is accurate. The study site may be subject to review by the Institutional Review Board (IRB) and/or appropriate regulatory authorities.

A CRF will be completed for each included subject and will be signed by the investigator or by an authorized staff member to attest that the data is true. Any corrections to entries made in the CRFs, source documents must be dated, initialed and explained (if necessary) and should not obscure the original entry. Qualit assurance will as also be performed regularly on the CRFs.

The primary end point will be analyzed using Time to event (cure, death, relapse etc)analysis and failure rates and hazard ratios will be calculated accordig to categorical drug concentrations with proposed cutt offs.

Secondary end points will be analysed using time to event for occurence of toxicities which will also be corelated to the drug concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Age of ≥18 years
* First episode of pulmonary TB i.e. proven or highly suspected TB considered for TB treatment qualifying for 6 months anti-Tb drugs regimen
* Confirmed HIV-1 infection

Exclusion Criteria:

* Unable to provide informed consent
* Documented or highly suspected TB infection of any organs/systems other than the lung requiring TB treatment longer than 6 months
* Previously treated for a mycobacterial infection (TB or atypical mycobacterial infection, active or latent)
* Pregnancy or planned pregnancy within the next year
* Unwillingness to perform pregnancy test
* Decompensated liver disease and/or aminotransferases >5x ULN
* GFR < 50 ml/min
* Co-morbidities reducing life expectancy to <1 year (e.g. cancer)
* Patient wishes to take part in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2013-02; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
clinical outcome | At the end of treatment (6 months after enrolmet)
  To investigate the association between serum concentrations of antituberculosis drugs and tuberculosis treatment response in HIV-TB-co-infected individuals.

SECONDARY OUTCOMES:
Cmax | At 2 weeks, 8 weeks and 24 weeks after anti-tuberculosis drug initiation
  To investigate the steady-state pharmacokinetic parameters of anti-TB drugs at different time-points over the course of TB-treatment
Number of adverse events | 2 weeks, 8 weeks and 24 weeks after anti-tuberculosis drug initiation
  To assess the safety and tolerability of anti-TB drugs based on the WHO guidelines
ART trough levels | At 2 weeks, 8 weeks and 24 weeks after anti-tuberculosis drug initiation
  To correlate the effect of anti-TB drugs on plasma concentrations of efavirenz or protease inhibitors and vice versa.
Isoniazid Cmax | At 2 weeks, 8 weeks and 24 weeks
  To evaluate the effect of acetylator geno-and phenotype (NAT-2 gene) on isoniazid plasma concentrations and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Castelnuovo, MD, PhD, Principal Investigator — Infectious Diseases Institute
Locations (1):
- Infectious Diseases Institute, Kampala, Kampala, Uganda

REFERENCES:
- [Background] Chideya S, Winston CA, Peloquin CA, Bradford WZ, Hopewell PC, Wells CD, Reingold AL, Kenyon TA, Moeti TL, Tappero JW. Isoniazid, rifampin, ethambutol, and pyrazinamide pharmacokinetics and treatment outcomes among a predominantly HIV-infected cohort of adults with tuberculosis from Botswana. Clin Infect Dis. 2009 Jun 15;48(12):1685-94. doi: 10.1086/599040. PMID 19432554
- [Background] Weiner M, Benator D, Burman W, Peloquin CA, Khan A, Vernon A, Jones B, Silva-Trigo C, Zhao Z, Hodge T; Tuberculosis Trials Consortium. Association between acquired rifamycin resistance and the pharmacokinetics of rifabutin and isoniazid among patients with HIV and tuberculosis. Clin Infect Dis. 2005 May 15;40(10):1481-91. doi: 10.1086/429321. Epub 2005 Apr 14. PMID 15844071
- [Background] Gurumurthy P, Ramachandran G, Hemanth Kumar AK, Rajasekaran S, Padmapriyadarsini C, Swaminathan S, Bhagavathy S, Venkatesan P, Sekar L, Mahilmaran A, Ravichandran N, Paramesh P. Decreased bioavailability of rifampin and other antituberculosis drugs in patients with advanced human immunodeficiency virus disease. Antimicrob Agents Chemother. 2004 Nov;48(11):4473-5. doi: 10.1128/AAC.48.11.4473-4475.2004. PMID 15504887
- [Background] Narita M, Hisada M, Thimmappa B, Stambaugh J, Ibrahim E, Hollender E, Ashkin D. Tuberculosis recurrence: multivariate analysis of serum levels of tuberculosis drugs, human immunodeficiency virus status, and other risk factors. Clin Infect Dis. 2001 Feb 1;32(3):515-7. doi: 10.1086/318490. Epub 2001 Jan 25. PMID 11170964
- [Background] Gumbo T, Louie A, Deziel MR, Liu W, Parsons LM, Salfinger M, Drusano GL. Concentration-dependent Mycobacterium tuberculosis killing and prevention of resistance by rifampin. Antimicrob Agents Chemother. 2007 Nov;51(11):3781-8. doi: 10.1128/AAC.01533-06. Epub 2007 Aug 27. PMID 17724157
- [Derived] Sekaggya-Wiltshire C, Chirehwa M, Musaazi J, von Braun A, Buzibye A, Muller D, Gutteck U, Motta I, Calcagno A, Fehr JS, Kambugu A, Castelnuovo B, Lamorde M, Denti P. Low Antituberculosis Drug Concentrations in HIV-Tuberculosis-Coinfected Adults with Low Body Weight: Is It Time To Update Dosing Guidelines? Antimicrob Agents Chemother. 2019 May 24;63(6):e02174-18. doi: 10.1128/AAC.02174-18. Print 2019 Jun. PMID 30910890
- [Derived] Sekaggya-Wiltshire C, von Braun A, Lamorde M, Ledergerber B, Buzibye A, Henning L, Musaazi J, Gutteck U, Denti P, de Kock M, Jetter A, Byakika-Kibwika P, Eberhard N, Matovu J, Joloba M, Muller D, Manabe YC, Kamya MR, Corti N, Kambugu A, Castelnuovo B, Fehr JS. Delayed Sputum Culture Conversion in Tuberculosis-Human Immunodeficiency Virus-Coinfected Patients With Low Isoniazid and Rifampicin Concentrations. Clin Infect Dis. 2018 Aug 16;67(5):708-716. doi: 10.1093/cid/ciy179. PMID 29514175
- [Derived] Kwizera R, Parkes-Ratanshi R, Page ID, Sekaggya-Wiltshire C, Musaazi J, Fehr J, Castelnuovo B, Kambugu A, Denning DW. Elevated Aspergillus-specific antibody levels among HIV infected Ugandans with pulmonary tuberculosis. BMC Pulm Med. 2017 Nov 21;17(1):149. doi: 10.1186/s12890-017-0500-9. PMID 29162063
- [Derived] Sekaggya-Wiltshire C, Castelnuovo B, von Braun A, Musaazi J, Muller D, Buzibye A, Gutteck U, Henning L, Ledergerber B, Corti N, Lamorde M, Fehr J, Kambugu A. Cohort profile of a study on outcomes related to tuberculosis and antiretroviral drug concentrations in Uganda: design, methods and patient characteristics of the SOUTH study. BMJ Open. 2017 Sep 18;7(9):e014679. doi: 10.1136/bmjopen-2016-014679. PMID 28928173